CLINICAL TRIAL: NCT03744442
Title: Efficacy of a Personalized Modular Intervention to Promote Dignity, Meaningfulness and Mindfulness by a Palliative Care Consultation-Liaison Service in Swiss Acute Hospital Care. A Feasibility Study
Brief Title: Promoting Dignity, Meaningfulness and Mental Well-Being
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Collaborators: Stanley Thomas Johnson Stiftung (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2018-01998, va18Eckstein
Record Dates: First submitted 2018-11-07; First posted 2018-11-16 (Actual); Last update posted 2024-04-11 (Actual); Status verified 2024-04

CONDITIONS: Life-limiting Serious Illness
Keywords: CALM Therapy; Dignity Therapy; Mindfulness-based intervention; Personalized Modular Intervention
MeSH Terms: interventions — Dignity Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Dignity Therapy (DT) module (Active Comparator): psychotherapeutic intervention asking patients about their most important achievements, roles and other important aspects of life; two structured sessions of 60 minutes conducted by a trained therapist
  Interventions: Procedure: Dignity Therapy (DT) module
- CALM Therapy module (Active Comparator): supportive-expressive psychotherapy aiming to help (1) manage the disease, symptom and treatment, and communicate with healthcare providers, to (2) adjust to changes in self-concept, personal relationships, and support needs, to (3) find a sense of meaning and purpose in life, and to (4) prepare for the future, sustain hope, and face the end of life; two structured sessions of 60 minutes conducted by a trained therapist
  Interventions: Procedure: CALM Therapy module
- Mindfulness-based interventions module (Active Comparator): Mind-body techniques reducing existential and spiritual distress and dealing with common experiences related to life-limiting diseases, including loss of control, uncertainty about the future; two structured sessions of 60 minutes conducted by a trained therapist
  Interventions: Procedure: Mindfulness-based interventions module

INTERVENTIONS:
Procedure: Dignity Therapy (DT) module — psychotherapeutic intervention asking patients about their most important achievements, roles and other important aspects of life; two structured sessions of 60 minutes conducted by a trained therapist
  Arms: Dignity Therapy (DT) module
Procedure: CALM Therapy module — supportive-expressive psychotherapy aiming to help (1) manage the disease, symptom and treatment, and communicate with healthcare providers, to (2) adjust to changes in self-concept, personal relationships, and support needs, to (3) find a sense of meaning and purpose in life, and to (4) prepare for the future, sustain hope, and face the end of life; two structured sessions of 60 minutes conducted by a trained therapist
  Arms: CALM Therapy module
Procedure: Mindfulness-based interventions module — Mind-body techniques reducing existential and spiritual distress and dealing with common experiences related to life-limiting diseases, including loss of control, uncertainty about the future; two structured sessions of 60 minutes conducted by a trained therapist
  Arms: Mindfulness-based interventions module

SUMMARY:
Feasibility study to test the feasibility and acceptability of a designed personalized modular Intervention consisting of three modules, including Cancer and Living Meaningfully (CALM) Therapy, Dignity Therapy (DT), and a mindfulness-based Intervention

DETAILED DESCRIPTION:
Patient with a life-limiting serious illness commonly experience substantial emotional and spiritual distress, death anxieties, depressive symptoms and loss of dignity and purpose in life. Fostering dignity and meaning and relieving psychological distress have been identified as a core objective for end-of-life care. However, individual's needs for dignity and psychological support at the end of life may vary. Therefore, a personalized approach is needed. On the basis of theoretical frameworks and existing dignity- fostering and meaning- based interventions, as well as an one-day workshop with international experts in the field of palliative care, a personalized modular intervention, consisting of three modules, including CALM Therapy, Dignity Therapy, and a mindfulness-based Intervention, was developed.

ELIGIBILITY:
Inclusion Criteria:

* Informed Consent as documented by signature
* Patients in palliative situation (i.e. patients suffering from an advanced, incurable, life-limiting disease with multimodal support needs)
* Estimated life expectancy ≤ 18 months
* Patients seen by the palliative consultation-liaison service at the University Hospital Basel as an in- or outpatient
* Willingness and capacity to commit at least three contacts over about 7-10 days

Exclusion Criteria:

* Being delirious or otherwise substantially cognitively impaired (based on clinical consensus)
* Being too ill to complete the requirements of the study protocol
* Unable to understand and speak German

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2020-03-05 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2023-11-15 (Actual)

PRIMARY OUTCOMES:
Change in acceptability of the personalized modular Intervention (motivation, satisfaction with Intervention, further recommendation) | baseline until 1-month follow- up
  Motivation for participating in the study, Satisfaction with the intervention, and If intervention would be recommended to other patients, measured by a semi-structured interview; assessment at baseline (T0), after the completion of the intervention (T1 = 2 weeks after baseline) and at 1-month follow- up (T2)
Rate of eligibility | at baseline (T0)
  feasibility of the personalized modular Intervention measured by rate of eligibility
Rate of consent | at baseline (T0)
  feasibility of the personalized modular Intervention measured by rate of consent
Final recruitment rate | at baseline (T0)
  feasibility of the personalized modular Intervention measured by final recruitment rate
Change in Patient adherence | baseline until 1-month follow- up
  feasibility of the personalized modular Intervention measured by rate of drop- Outs; assessment at baseline (T0), after the completion of the intervention (T1 = 2 weeks after baseline) and at 1-month follow- up (T2)
Change in Questionnaire completion rates | baseline until 1-month follow- up
  feasibility of the personalized modular Intervention measured by rate of completion of questionnaire and expenditure of time for completing questionnaire (in minutes); assessment at baseline (T0), after the completion of the intervention (T1 = 2 weeks after baseline) and at 1-month follow- up (T2)

SECONDARY OUTCOMES:
Change in Patient Health Questionnaire-9 (PHQ-9) | baseline until 1-month follow- up
  PHQ-9 is a 9-question instrument given to patients to screen for the presence and severity of Depression. Scores Depression severity from 0 (=none) to 27 (severe); assessment at baseline (T0), after the completion of the intervention (T1 = 2 weeks after baseline) and at 1-month follow- up (T2)
Change in Patient Dignity Inventory (PDI) | baseline until 1-month follow- up
  25-item PDI measurement of various sources of dignity-related distress among patients nearing the end of life; each item rated on a five-point scale (1=not a problem; 2= a slight problem; 3=a problem; 4=a major problem; 5=an overwhelming problem); assessment at baseline (T0), after the completion of the intervention (T1 = 2 weeks after baseline) and at 1-month follow- up (T2)
Change in Death and Dying Distress Scale (DADDS) | baseline until 1-month follow- up
  15-item scale to assess concerns related to death and dying in patients with advanced cancer. Items are answered on a 6-point scale from 0 (no distress) to 5 (extreme distress). Total scores may range from 0 to 75 and scores ≥45 refer to the presence of at least moderate death anxiety. Assessment at baseline (T0), after the completion of the intervention (T1 = 2 weeks after baseline) and at 1-month follow- up (T2)

CONTACTS AND LOCATIONS:
Overall Officials: Sandra Eckstein, Dr. med, Principal Investigator — Department of Psychosomatic Medicine, University Hospital Basel
Locations (1):
- Department of Psychosomatics, University Hospital of Basel, Basel, Switzerland